CLINICAL TRIAL: NCT04784000
Title: A Phase 1 Study Assessing the Effect of Carbamazepine, a P-Glycoprotein Inducer, on the Pharmacokinetics of AT-527 in Healthy Adult Subjects
Brief Title: Effect of Carbamazepine on the Pharmacokinetics (PK) of AT-527
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-004
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT-527 550 mg + carbamezepine (Experimental)
  Interventions: Drug: Period 1: AT-527 550 mg; Drug: Period 2: carbamazepine; Drug: Period 3: AT-527 550 mg + carbamazepine
- AT-527 1100 mg + carbamezepine (Experimental)
  Interventions: Drug: Period 1: AT-527 550 mg; Drug: Period 2: carbamazepine; Drug: Period 3: AT-527 1100 mg + carbamazepine

INTERVENTIONS:
Drug: Period 1: AT-527 550 mg — AT-527 550 mg tablet (1 x 550 mg tablet, in the morning) on Day 1
  Other Names: AT-527 is also known as RO7496998
Drug: Period 2: carbamazepine — Carbamazepine 100 mg twice daily (BID) Days 3 to 6, 200 mg BID on Days 9 to 11, 300 mg BID on Days 12 to 25
Drug: Period 3: AT-527 550 mg + carbamazepine — AT-527 550 mg tablet (1 x 550 mg tablet, in the morning) on Day 26 plus carbamazepine 300 mg BID on Day 26
  Other Names: AT-527 is also known as RO7496998
  Arms: AT-527 550 mg + carbamezepine
Drug: Period 3: AT-527 1100 mg + carbamazepine — AT-527 1100 mg tablet (2 x 550 mg tablets, in the morning) on Day 26 plus carbamazepine 300 mg BID on Day 26
  Other Names: AT-527 is also known as RO7496998
  Arms: AT-527 1100 mg + carbamezepine

SUMMARY:
This study will determine the effect of carbamazepine on the PK of AT-527 (RO7496998) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-29 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus, hepatitis C virus, HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Use of other prescription drugs with 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of AT-527 (RO7496998) | Day 1 vs Day 26
  Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) of AT-527 (RO7496998) | Day 1 vs Day 26
  Area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Montreal, Quebec, Canada